CLINICAL TRIAL: NCT02462356
Title: A Randomized Controlled Study: the Effect of Multiple-portal VATS Versus Conventional VATS Lobectomy for NSCLC
Brief Title: Multiple-portal VATS Versus Uniportal VATS Lobectomy for Non-small Cell Lung Cancer
Acronym: MVUVLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Junqiang Fan, Thoracic Surgery Department, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY15H160034
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: CVATS; UVATS; perioperative effect; ergonomic influence
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional VATS (Active Comparator): Via conventional VATS lobectomy and systematic lymph node dissection for lung cancer
  Interventions: Procedure: Conventional VATS
- Uniportal VATS (Experimental): Via uniportal VATS lobectomy and systematic lymph node dissection for lung cancer
  Interventions: Procedure: Uniportal VATS

INTERVENTIONS:
Procedure: Uniportal VATS — Uniportal VATS lobectomy and lymph node dissection will be performed in this group
  Arms: Uniportal VATS
Procedure: Conventional VATS — Conventional VATS lobectomy and lymph node dissection will be performed in this group
  Arms: Conventional VATS

SUMMARY:
This study evaluate multiple-portal VATS and uniportal VATS lobectomy for NSCLC, half of participants will receive multiple VATS, while the other half will receive uniportal VATS lobectomy.

DETAILED DESCRIPTION:
Conventional VATS and uniportal VATS lobectomy can be performed each for NSCLC. Conventional VATS lobectomy employ 3 or 4 ports for completing the operation. Usually the camera port is performed at the seventh or eighth intercostals space within the trocar, so it's easy to cause the intercostals nerve and vessel injure, and still create obvious pain.

However, the lobectomy for lung cancer can be accomplished with a single incision. According to the initial results, Uniportal VATS (UVATS) lobectomy procedure has been wide adopted by less acess trauma, relieve postoperative pain. But these were retrospective and descriptive, not randomized study. Further randomized control studies will be required to demonstrate that there are more benefits in UVATS techniques compared with conventional VATS for lobectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of primary lung cancer with the age between 35 and 75 years old;
* Patients with Tumor size ≤5cm，clinically staged T1-2N0-1M0，prepared for lobectomy and mediastinal lymph node dissection;
* Patients with an American Society of Anesthesiology score of 0-1.

Exclusion Criteria:

* Patients with N2 or N3 positive or distant metastasis.
* Patients who had undergone Neoadjuvant chemotherapy.
* Patients with tumor invasion to the peripheral structures.
* Patients with previous history of thoracic operations.
* Patients with serious thoracic adhesion.
* Patients who will undergo Pneumonectomy, sleeve lobectomy, segmentectomy, wedge resection.
* Patients with preexisting chronic obstructive pulmonarydisease, asthma, or interstitial lung disease;
* Patients with cardiac, hepatic, or renal dysfunction;

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
short-term quality of life(EQ5D) between the two groups | Up to 6 month
  To observe differences of short-term effects(bleeding volume during operation,operation time, hospital mortality, hospital stay and so on) between two groups.

SECONDARY OUTCOMES:
intra-operative and postoperative complications | form the day of surgery up to discharege (expected within 1 month)
  Surgical Complications include conversion rate, bleeding, air leakage, pain, cardiac arrhythmias, wound infection, pulmonary complications, pulmonary function will be measured.
lung function | pre-operative, 3 weeks, 3 months after surgery
  lung function will be measured at pre-operative, 3 weeks, 3 months after surgery
Pain Scores after surgery | 1, 3 days and 1, 3 months after surgery
  Pain Scores will be measured by Brief pain inventory
The surgeon's ergonomic influence during operation(blinks/min) | The video is capture every 5 minutes and lasted for 1 minute
  Spontaneous eye blink rate(NASA Task Load Index，NASA TLX)

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital Zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yao J, Chang Z, Zhu L, Fan J. Uniportal versus multiportal thoracoscopic lobectomy: Ergonomic evaluation and perioperative outcomes from a randomized and controlled trial. Medicine (Baltimore). 2020 Oct 16;99(42):e22719. doi: 10.1097/MD.0000000000022719. PMID 33080728